CLINICAL TRIAL: NCT07331961
Title: Assessment of the Feasibility and Clinical Efficacy of Low-Intensity Extracorporeal Shockwave Therapy (Li-ESWT) Using the Dornier System in Patients With Vasculogenic Erectile Dysfunction: A Pilot Study
Brief Title: The Feasibility of Using Dornier Machine in Patients With Erectile Dysfunction, a Pilot Study.
Acronym: DED-Pilot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelrahman Mohamed Abdelkader, teaching assistant, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESWT in erectile dysfunction
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Erectile Dysfunction (ED)
Keywords: erectile dysfunction; low intensity shock wave treatment; extracorporeal shock wave therapy
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- patients diagnosed with erectile dysfunctiom (Experimental): they will receive shock wave therapy on their penis by using a machine that is not designed for this purpose.
  Interventions: Device: extracorporeal shock wave therpy

INTERVENTIONS:
Device: extracorporeal shock wave therpy — we will use a Dornier lithotripsy delta 2 for treatment of patient with erectile dysfunction

SUMMARY:
Extracorporeal Shockwave Therapy (ESWT) is a well-established modality for treating various urological and musculoskeletal conditions. Recently, its application has expanded to include vasculogenic erectile dysfunction (ED), primarily due to its ability to trigger neo-angiogenesis and significantly improve penile blood flow.

DETAILED DESCRIPTION:
Extracorporeal Shockwave Therapy (ESWT) is a well-established modality for treating various urological and musculoskeletal conditions. Recently, its application has expanded to include vasculogenic erectile dysfunction (ED), primarily due to its ability to trigger neo-angiogenesis and significantly improve penile blood flow. While the clinical efficacy of Low-Intensity Extracorporeal Shockwave Therapy (Li-ESWT) is increasingly recognized globally, it currently remains non-FDA approved for this specific indication. Furthermore, the accessibility of this treatment is often limited, as dedicated Li-ESWT machines are expensive and frequently unavailable in public healthcare settings.

This pilot study investigates the feasibility of adapting the Dornier Delta Lithotripter utilized for high-energy renal stone fragmentation for penile therapy. The central research question focuses on whether this high-energy platform can be safely and precisely calibrated to low-intensity levels to provide therapeutic benefits without inducing tissue damage and complications.

Our clinical rationale is inspired by shifting paradigms in other medical fields, such as prostate cancer radiotherapy, which emphasize delivering a concentrated therapeutic dose in fewer sessions. Since early pilot studies most notably by Vardi et al experimented with standardized five-point techniques over multiple weeks, we seek to optimize this by evaluating the impact of focused energy delivery and modified patient positioning.This research aims to provide a cost-effective, accessible alternative for ED treatment using existing hospital infrastructure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with erectile dysfunction (ED) confirmed by clinical assessment and penile duplex Doppler ultrasound

Exclusion Criteria:

* 1-Coagulapathy. 2-Penile prosthesis. 3-Post Radical Cystectomy 4-Intellectual disability 5-Skeletal abnormalty

Min Age: 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — males
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
detection of complications from the use of ESWL machine | follow up will begin after the first session and then repeated weekly for 1 month
  the patients will be evaluated after the procedure for 1 month to identify any side-effects as hematoma or difficult urination
improvement in the international erectile function score | follow up will begin after day one and then repeated weekly for 1 month

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Result] Rosen RC, Allen KR, Ni X, Araujo AB. Minimal clinically important differences in the erectile function domain of the International Index of Erectile Function scale. Eur Urol. 2011 Nov;60(5):1010-6. doi: 10.1016/j.eururo.2011.07.053. Epub 2011 Jul 30. PMID 21855209
- [Result] Ergun O, Kim K, Kim MH, Hwang EC, Blair Y, Gudeloglu A, Parekattil S, Dahm P. Low-intensity shockwave therapy for erectile dysfunction. Cochrane Database Syst Rev. 2025 Jul 14;7(7):CD013166. doi: 10.1002/14651858.CD013166.pub3. PMID 40654049
- [Result] Vardi Y, Appel B, Jacob G, Massarwi O, Gruenwald I. Can low-intensity extracorporeal shockwave therapy improve erectile function? A 6-month follow-up pilot study in patients with organic erectile dysfunction. Eur Urol. 2010 Aug;58(2):243-8. doi: 10.1016/j.eururo.2010.04.004. Epub 2010 May 6. PMID 20451317
- [Result] Kalyvianakis D, Mykoniatis I, Pyrgidis N, Kapoteli P, Zilotis F, Fournaraki A, Hatzichristou D. The Effect of Low-Intensity Shock Wave Therapy on Moderate Erectile Dysfunction: A Double-Blind, Randomized, Sham-Controlled Clinical Trial. J Urol. 2022 Aug;208(2):388-395. doi: 10.1097/JU.0000000000002684. Epub 2022 May 6. PMID 35830338